CLINICAL TRIAL: NCT01466790
Title: An Exploratory Phase IIa, Randomized, Open-Label Trial to Investigate the Efficacy and Safety of 12 Weeks or 24 Weeks of TMC435 in Combination With PSI-7977 (GS7977) With Or Without Ribavirin in Chronic Hepatitis C Genotype 1-Infected Prior Null Responders To Peginterferon/Ribavirin Therapy or HCV Treatment-Naive Subjects
Brief Title: A Study of TMC435 in Combination With PSI-7977 (GS7977) in Chronic Hepatitis C Genotype 1-Infected Prior Null Responders To Peginterferon/Ribavirin Therapy or HCV Treatment-Naive Patients
Acronym: COSMOS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR018724; TMC435HPC2002 (Other: Janssen R&D Ireland)
Record Dates: First submitted 2011-11-03; First posted 2011-11-08 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2015-02-09 (Estimated); Status verified 2015-01

CONDITIONS: Hepatitis C
Keywords: Hepatitis C; TMC435; PSI-7977; GS7977; Ribavirin; HCV; Hep C; Genotype 1
MeSH Terms: conditions — Hepatitis C | interventions — Simeprevir; Sofosbuvir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm 1 (Experimental): 30 patients will receive TMC435 (150 mg once a day) plus PSI-7977(GS7977) (400 mg once a day) with ribavirin (1000-1200 mg/day) for 24 weeks and followed by a 24-week follow-up phase.
  Interventions: Drug: TMC435; Drug: PSI-7977 (GS7977); Drug: Ribavirin
- Arm 2 (Experimental): 15 patients wiil receive TMC435 (150 mg once a day) plus PSI-7977 (GS7977) (400 mg once a day) for 24 weeks of and followed by a 24-week follow-up phase.
  Interventions: Drug: TMC435; Drug: PSI-7977 (GS7977)
- Arm 3 (Experimental): 30 patients will receive TMC435 (150 mg once a day) plus PSI-7977 (GS7977) (400 mg once a day) with ribavirin (1000-1200 mg/day) for 12 weeks and followed by a 36-week follow-up phase.
  Interventions: Drug: TMC435; Drug: PSI-7977 (GS7977); Drug: Ribavirin
- Arm 4 (Experimental): 15 patients will receive TMC435 (150 mg once a day) plus PSI-7977 (GS7977) (400 mg once a day) for 12 weeks and followed by a 36-week follow-up phase.
  Interventions: Drug: TMC435; Drug: PSI-7977 (GS7977)

INTERVENTIONS:
Drug: TMC435 — TMC435 will be administered as one oral capsule of 150 mg once a day.
Drug: PSI-7977 (GS7977) — PSI-7977 (GS7977) will be administered as oral tablets (2 tablets of 200 mg for Cohort 1 and 1 tablet of 400 mg for Cohort 2) once a day.
  Other Names: GS7977
Drug: Ribavirin — Ribavirin will be administered according to body weight. For patients with body weight less than 75 kg daily dose (1000 mg) will be administered as 400 mg (2 oral tablets of 200 mg) in the morning and 600 mg (3 oral tablets of 200 mg) in the evening. Body weight more than or equal to 75 kg daily dose (1200 mg) will be administered as 600 mg twice a day (3 tablets of 200 mg per intake, morning and evening).
  Arms: Arm 1; Arm 3

SUMMARY:
The purpose of this study is to investigate the efficacy and safety of TMC435 plus PSI-7977 (GS7977) with or without ribavirin in patients who are chronically infected with genotype 1 hepatitis C virus (HCV) and who did not respond to prior peginterferon/ribavirin therapy or are HCV treatment-naive (patients who never received treatment for HCV infection).

DETAILED DESCRIPTION:
This is a Phase IIa, randomized (the study medications are assigned by chance), open label (all people know the identity of the intervention) study of TMC435 plus PSI-7977 (GS7977) with or without ribavirin. The study consists of a screening phase (6 weeks); a treatment phase (12 or 24 week period); and a posttreatment phase (follow-up period up to Week 48). Approximately 180 patients will be enrolled in this study. Patients will be sequentially enrolled into two cohorts in this study. Cohort 1 (90 patients) will include patients without advanced hepatic fibrosis who did not respond to previous PegIFN/ribavirin therapy and Cohort 2 (90 patients) will include only patients with advanced hepatic fibrosis who did not respond to previous PegIFN/ribavirin therapy or are HCV treatment-naive. Safety will be evaluated throughout the study and will include evaluations of adverse events, clinical laboratory tests, electrocardiogram, vital signs, and physical examination. The entire study duration for each participant will be approximately 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Chronic genotype 1 hepatitis C virus (HCV) infection
* Plasma HCV RNA of more than 10,000 IU/mL at screening
* Patients in Cohort 1 must be null responders to PegIFN/ribavirin with at least 1 documented previous course of PegIFN/ribavirin therapy for at least 12 consecutive weeks
* Patients in Cohort 2 must be null responders to PegIFN/ribavirin with at least 1 documented previous course of PegIFN/ribavirin therapy for at least 12 consecutive weeks and could also be HCV treatment-naive, meaning never received treatment with any approved or investigational drug for the treatment of HCV
* Null responders patients in Cohort 1 and Cohort 2 must meet the defined criterion for a null responder, defined as on-treatment less than 2 log10 IU/mL reduction in HCV RNA from baseline at Week 12 of the most recent PegIFN/ribavirin therapy
* Patient must have had a liver biopsy within 3 years before screening (or between screening and baseline visit) or patient must have had a liver biopsy at any time in the past which showed Metavir F3 or F4 fibrosis
* Must agree to use 2 forms of effective contraception throughout the study (male and female)

Exclusion Criteria:

* Has evidence of hepatic decompensation
* Has any liver disease of non-HCV etiology
* Has an infection/co-infection with non-genotype 1 HCV
* Has a co-infection with Human immunodeficiency virus (HIV) type 1 or type 2 (HIV-1 or HIV-2) (positive HIV-1 or HIV-2 antibody test at screening)
* Has a co-infection with hepatitis B virus (hepatitis B surface antigen [HBsAg] positive)
* Has a history of malignancy within 5 years of the screening visit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2012-01; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (23):
- United States (22):
  - Hoover, Alabama
  - Bakersfield, California
  - La Jolla, California
  - San Diego, California
  - New Haven, Connecticut
  - Brandenton, Florida
  - Jacksonville, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Wellington, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Lutherville, Maryland
  - Lebanon, New Hampshire
  - New York, New York
  - Pittsburgh, Pennsylvania
  - Arlington, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Falls Church, Virginia
  - Norfolk, Virginia
  - Seatle, Washington
- Santurce, Puerto Rico

REFERENCES:
- [Derived] Lawitz E, Sulkowski MS, Ghalib R, Rodriguez-Torres M, Younossi ZM, Corregidor A, DeJesus E, Pearlman B, Rabinovitz M, Gitlin N, Lim JK, Pockros PJ, Scott JD, Fevery B, Lambrecht T, Ouwerkerk-Mahadevan S, Callewaert K, Symonds WT, Picchio G, Lindsay KL, Beumont M, Jacobson IM. Simeprevir plus sofosbuvir, with or without ribavirin, to treat chronic infection with hepatitis C virus genotype 1 in non-responders to pegylated interferon and ribavirin and treatment-naive patients: the COSMOS randomised study. Lancet. 2014 Nov 15;384(9956):1756-65. doi: 10.1016/S0140-6736(14)61036-9. Epub 2014 Jul 28. PMID 25078309

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 168 participants enrolled to study. 1 participant who was randomized to Cohort 1: TMC435, PSI-7977 and Ribavirin for 24 Weeks group, but never received treatment.
Groups:
- Cohort 1: TMC435, PSI-7977 and Ribavirin for 24 Weeks: Cohort 1 participants (without advanced hepatic fibrosis, who did not respond to previous pegylated interferon [PegIFN]/ribavirin therapy) received TMC435 150 milligram (mg) capsule along with PSI-7977 (GS7977) 400 mg tablet and ribavirin 1000-1200 mg tablet (1000 mg for participants with body weight less than 75 kilogram [kg] and 1200 mg for participants with body weight more than or equal to 75 kg) orally once daily for 24 weeks followed by a 24-week follow-up phase.
- Cohort 1: TMC435 and PSI-7977 for 24 Weeks: Cohort 1 participants received TMC435 150 mg capsule along with PSI-7977 (GS7977) 400 mg tablet orally once daily for 24 weeks followed by a 24-week follow-up phase.
- Cohort 1: TMC435, PSI-7977 and Ribavirin for 12 Weeks: Cohort 1 participants received TMC435 150 mg capsule along with PSI-7977 (GS7977) 400 mg tablet and ribavirin 1000-1200 mg tablet (1000 mg for participants with body weight less than 75 kg and 1200 mg for participants with body weight more than or equal to 75 kg) orally once daily for 12 weeks followed by a 36-week follow-up phase.
- Cohort 1: TMC435 and PSI-7977 for 12 Weeks: Cohort 1 participants received TMC435 150 mg capsule along with PSI-7977 (GS7977) 400 mg tablet orally once daily for 12 weeks followed by a 36-week follow-up phase.
- Cohort 2: TMC435, PSI-7977 and Ribavirin for 24 Weeks: Cohort 2 participants (with advanced hepatic fibrosis, who did not respond to previous PegIFN/ribavirin therapy or who never received treatment for HCV infection) received TMC435 150 mg capsule along with PSI-7977 400 mg tablet and ribavirin 1000-1200 mg tablet (1000 mg for participants with body weight less than 75 kg and 1200 mg for participants with body weight more than or equal to 75 kg) orally once daily for 24 weeks followed by a 24-week follow-up phase.
- Cohort 2: TMC435 and PSI-7977 for 24 Weeks: Cohort 2 participants received TMC435 150 mg capsule along with PSI-7977 400 mg tablet orally once daily for 24 weeks followed by a 24-week follow-up phase.
- Cohort 2: TMC435, PSI-7977 and Ribavirin for 12 Weeks: Cohort 2 participants received TMC435 150 mg capsule along with PSI-7977 400 mg tablet and ribavirin 1000-1200 mg tablet (1000 mg for participants with body weight less than 75 kg and 1200 mg for participants with body weight more than or equal to 75 kg) orally once daily for 12 weeks followed by a 36-week follow-up phase.
- Cohort 2: TMC435 and PSI-7977 for 12 Weeks: Cohort 2 participants received TMC435 150 mg capsule along with PSI-7977 400 mg tablet orally once daily for 12 weeks followed by a 36-week follow-up phase.
Period: Overall Study
Arm/Group | Cohort 1: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 1: TMC435 and PSI-7977 for 24 Weeks | Cohort 1: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 1: TMC435 and PSI-7977 for 12 Weeks | Cohort 2: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 2: TMC435 and PSI-7977 for 24 Weeks | Cohort 2: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 2: TMC435 and PSI-7977 for 12 Weeks
Started | 24 (Not including 1 participant who was randomized to this group, but never received treatment.) | 15 | 27 | 14 | 30 | 16 | 27 | 14
Completed | 20 | 14 | 27 | 14 | 27 | 16 | 26 | 13
Not Completed | 4 | 1 | 0 | 0 | 3 | 0 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 1: TMC435 and PSI-7977 for 24 Weeks | Cohort 1: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 1: TMC435 and PSI-7977 for 12 Weeks | Cohort 2: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 2: TMC435 and PSI-7977 for 24 Weeks | Cohort 2: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 2: TMC435 and PSI-7977 for 12 Weeks | Total
Number analyzed (Participants) | 24 | 15 | 27 | 14 | 30 | 16 | 27 | 14 | 167
Age, Continuous [Median (Full Range); unit: years] | 56 [27 to 70] | 56 [27 to 61] | 55 [28 to 67] | 55.5 [35 to 68] | 58 [28 to 70] | 57.5 [49 to 63] | 57 [36 to 68] | 57.5 [47 to 64] | 57 [27 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 7 | 6 | 9 | 9 | 7 | 4 | 60
  Male | 15 | 6 | 20 | 8 | 21 | 7 | 20 | 10 | 107

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Sustained Virologic Response (SVR) 12 Weeks After the Planned End of Treatment (EOT)
Description: Participants with hepatitis C virus (HCV) ribonucleic acid (RNA) undetectable at end of treatment and HCV RNA less than (<) 25 international unit per milliliter (IU/mL) (detectable or undetectable) at 12 weeks after the planned end of treatment.
Time Frame: Week 12 and 24 (for the arms treated for 12 weeks) or Week 24 and 36 (for the arms treated for 24 weeks)
Population: Intention-to-treat (ITT) population included all randomized participants who took at least one dose of investigational drug.
Measure: Number; unit: Participants
Arm/Group | Cohort 1: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 1: TMC435 and PSI-7977 for 24 Weeks | Cohort 1: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 1: TMC435 and PSI-7977 for 12 Weeks | Cohort 2: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 2: TMC435 and PSI-7977 for 24 Weeks | Cohort 2: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 2: TMC435 and PSI-7977 for 12 Weeks
Number analyzed (Participants) | 24 | 15 | 27 | 14 | 30 | 16 | 27 | 14
Participants | 19 | 14 | 26 | 13 | 28 | 16 | 25 | 13

2. Secondary Outcome: Number of Participants With a Sustained Virologic Response (SVR) 4 Weeks After the Planned End of Treatment (EOT)
Description: Participants with hepatitis C virus (HCV) ribonucleic acid (RNA) undetectable at end of treatment and HCV RNA less than (<) 25 international unit per milliliter (IU/mL) (detectable or undetectable) at 4 weeks after the planned end of treatment.
Time Frame: Week 12 and 16 (for the arms treated for 12 weeks) or Week 24 and 28 (for the arms treated for 24 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cohort 1: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 1: TMC435 and PSI-7977 for 24 Weeks | Cohort 1: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 1: TMC435 and PSI-7977 for 12 Weeks | Cohort 2: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 2: TMC435 and PSI-7977 for 24 Weeks | Cohort 2: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 2: TMC435 and PSI-7977 for 12 Weeks
Number analyzed (Participants) | 24 | 15 | 27 | 14 | 30 | 16 | 27 | 14
Participants | 20 | 14 | 26 | 13 | 28 | 16 | 26 | 14

3. Secondary Outcome: Number of Participants With a Sustained Virologic Response (SVR) 24 Weeks After the Planned End of Treatment (EOT)
Description: Participants with HCV RNA undetectable at end of treatment and HCV RNA less than (<) 25 IU/mL (detectable or undetectable) at 24 weeks after the planned end of treatment.
Time Frame: Week 12 and 36 (for the arms treated for 12 weeks) or Week 24 and 48 (for the arms treated for 24 weeks)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cohort 1: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 1: TMC435 and PSI-7977 for 24 Weeks | Cohort 1: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 1: TMC435 and PSI-7977 for 12 Weeks | Cohort 2: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 2: TMC435 and PSI-7977 for 24 Weeks | Cohort 2: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 2: TMC435 and PSI-7977 for 12 Weeks
Number analyzed (Participants) | 24 | 15 | 27 | 14 | 30 | 16 | 27 | 14
Participants | 19 | 14 | 26 | 13 | 28 | 16 | 25 | 13

4. Secondary Outcome: Number of Participants With a Sustained Virologic Response (SVR) at Week 48
Description: Participants with HCV RNA undetectable at end of treatment and HCV RNA less than (<) 25 IU/mL (detectable or undetectable) at week 48.
Time Frame: Week 48
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cohort 1: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 1: TMC435 and PSI-7977 for 24 Weeks | Cohort 1: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 1: TMC435 and PSI-7977 for 12 Weeks | Cohort 2: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 2: TMC435 and PSI-7977 for 24 Weeks | Cohort 2: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 2: TMC435 and PSI-7977 for 12 Weeks
Number analyzed (Participants) | 24 | 15 | 27 | 14 | 30 | 16 | 27 | 14
Participants | 19 | 14 | 26 | 13 | 27 | 16 | 24 | 13

5. Secondary Outcome: Number of Participants With Viral Breakthrough
Description: Viral breakthrough was defined as confirmed quantifiable HCV RNA after becoming less than (<) lower limit of quantification (LLOQ) or confirmed greater than (>) 1 log10 HCV RNA increase from the lowest level reached on 2 consecutive occasions.
Time Frame: Up to End of Treatment [Week 12 (for the arms treated for 12 weeks) or Week 24 (for the arms treated for 24 weeks)]
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cohort 1: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 1: TMC435 and PSI-7977 for 24 Weeks | Cohort 1: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 1: TMC435 and PSI-7977 for 12 Weeks | Cohort 2: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 2: TMC435 and PSI-7977 for 24 Weeks | Cohort 2: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 2: TMC435 and PSI-7977 for 12 Weeks
Number analyzed (Participants) | 24 | 15 | 27 | 14 | 30 | 16 | 27 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Inadequate Virologic Response
Description: Inadequate Virologic Response was defined as confirmed detectable HCV RNA at or after Week 8 and not meeting the viral breakthrough definition.
Time Frame: Week 8 and End of Treatment [Week 12 (for the arms treated for 12 weeks) or Week 24 (for the arms treated for 24 weeks)]
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cohort 1: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 1: TMC435 and PSI-7977 for 24 Weeks | Cohort 1: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 1: TMC435 and PSI-7977 for 12 Weeks | Cohort 2: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 2: TMC435 and PSI-7977 for 24 Weeks | Cohort 2: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 2: TMC435 and PSI-7977 for 12 Weeks
Number analyzed (Participants) | 24 | 15 | 27 | 14 | 30 | 16 | 27 | 14
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Viral Relapse
Description: Viral relapse was defined as undetectable HCV RNA at the actual EOT and confirmed quantifiable HCV RNA (>= 25 IU/mL) during follow-up period.
Time Frame: During the Follow-up [Week 36 (for the arms treated for 12 weeks) or Week 24 (for the arms treated for 24 weeks)]
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Cohort 1: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 1: TMC435 and PSI-7977 for 24 Weeks | Cohort 1: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 1: TMC435 and PSI-7977 for 12 Weeks | Cohort 2: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 2: TMC435 and PSI-7977 for 24 Weeks | Cohort 2: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 2: TMC435 and PSI-7977 for 12 Weeks
Number analyzed (Participants) | 24 | 15 | 27 | 14 | 30 | 16 | 27 | 14
Participants | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 1

ADVERSE EVENTS:
Time Frame: Up to Week 48
Groups:
- Cohort 1 and 2: TMC435, PSI-7977 and Ribavirin for 24 Weeks: Cohorts 1 and 2 participants received TMC435 150 mg capsule along with PSI-7977 400 mg tablet and ribavirin 1000-1200 mg tablet (1000 mg for participants with body weight less than 75 kg and 1200 mg for participants with body weight more than or equal to 75 kg) orally once daily for 24 weeks followed by a 24-week follow-up phase.
- Cohort 1 and 2: TMC435 and PSI-7977 for 24 Weeks: Cohorts 1 and 2 participants received TMC435 150 mg capsule along with PSI-7977 400 mg tablet orally once daily for 24 weeks followed by a 24-week follow-up phase.
- Cohort 1 and 2: TMC435, PSI-7977 and Ribavirin for 12 Weeks: Cohorts 1 and 2 participants received TMC435 150 mg capsule along with PSI-7977 400 mg tablet and ribavirin 1000-1200 mg tablet (1000 mg for participants with body weight less than 75 kg and 1200 mg for participants with body weight more than or equal to 75 kg) orally once daily for 12 weeks followed by a 36-week follow-up phase.
- Cohort 1 and 2: TMC435 and PSI-7977 for 12 Weeks: Cohorts 1 and 2 participants received TMC435 150 mg capsule along with PSI-7977 400 mg tablet orally once daily for 12 weeks followed by a 36-week follow-up phase.
Arm/Group | Cohort 1 and 2: TMC435, PSI-7977 and Ribavirin for 24 Weeks | Cohort 1 and 2: TMC435 and PSI-7977 for 24 Weeks | Cohort 1 and 2: TMC435, PSI-7977 and Ribavirin for 12 Weeks | Cohort 1 and 2: TMC435 and PSI-7977 for 12 Weeks
Serious Adverse Events (participants affected / at risk) | 3/54 | 1/31 | 0/54 | 0/28
Other Adverse Events (participants affected / at risk) | 48/54 | 25/31 | 42/54 | 17/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 and 2: TMC435, PSI-7977 and Ribavirin for 24 Weeks (N=54) | Cohort 1 and 2: TMC435 and PSI-7977 for 24 Weeks (N=31) | Cohort 1 and 2: TMC435, PSI-7977 and Ribavirin for 12 Weeks (N=54) | Cohort 1 and 2: TMC435 and PSI-7977 for 12 Weeks (N=28)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Retinal tear (Eye disorders) | 1 | 0 | 0 | 0
Visual impairment (Eye disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 and 2: TMC435, PSI-7977 and Ribavirin for 24 Weeks (N=54) | Cohort 1 and 2: TMC435 and PSI-7977 for 24 Weeks (N=31) | Cohort 1 and 2: TMC435, PSI-7977 and Ribavirin for 12 Weeks (N=54) | Cohort 1 and 2: TMC435 and PSI-7977 for 12 Weeks (N=28)
Anaemia (Blood and lymphatic system disorders) | 13 | 0 | 6 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 0 | 2 | 0
Constipation (Gastrointestinal disorders) | 4 | 1 | 4 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 5 | 3 | 2
Dry mouth (Gastrointestinal disorders) | 3 | 0 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 1 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 7 | 4 | 9 | 6
Toothache (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1 | 0
Chills (General disorders) | 3 | 0 | 1 | 0
Fatigue (General disorders) | 21 | 10 | 14 | 7
Influenza like illness (General disorders) | 1 | 2 | 0 | 0
Oedema peripheral (General disorders) | 4 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1 | 4 | 0
Seasonal allergy (Immune system disorders) | 3 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 2 | 2 | 0 | 0
Oral herpes (Infections and infestations) | 4 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 2 | 3 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 6 | 1
Urinary tract infection (Infections and infestations) | 3 | 2 | 1 | 0
Sunburn (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 2
Blood amylase increased (Investigations) | 2 | 2 | 4 | 0
Blood creatine phosphokinase increased (Investigations) | 4 | 2 | 6 | 1
Lipase increased (Investigations) | 2 | 1 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 3 | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2 | 2 | 0
Dizziness (Nervous system disorders) | 7 | 5 | 3 | 1
Headache (Nervous system disorders) | 11 | 7 | 9 | 6
Memory impairment (Nervous system disorders) | 1 | 2 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 0 | 0 | 3 | 1
Insomnia (Psychiatric disorders) | 9 | 2 | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 3 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 3 | 3 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 1 | 2 | 2
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 1 | 5 | 3
Rash (Skin and subcutaneous tissue disorders) | 7 | 3 | 8 | 1
Hypertension (Vascular disorders) | 2 | 2 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less